CLINICAL TRIAL: NCT02526550
Title: Immunogenicity of a Live Attenuated Chimeric Japanese Encephalitis Vaccine (IMOJEV) as a Booster Dose After a Primary Vaccination With CD.JEVAX in Thai Children
Brief Title: Immunogenicity of a Live Attenuated Chimeric JE Vaccine (IMOJEV) as a Booster Dose in Thai Children Primed With CD.JEVAX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Kulkanya Chokephaibulkit, Professor, Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JEC26-EXT
Record Dates: First submitted 2015-08-09; First posted 2015-08-18 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-10

CONDITIONS: Encephalitis
Keywords: Live attenuated Japanese Encephalitis vaccine; IMOJEV; CD.JEVAX; Booster; Thai children; Immunogenicity; Safety; Interchangeability; Hepatitis A vaccine; Vaccination or Other Immunization Procedure
MeSH Terms: conditions — Encephalitis; Hepatitis | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imojev (Experimental): Live attenuated chimeric Japanese Encephalitis vaccine, 0.5 mL dose containing ≥ 4.0 log10 plaque forming units (PFU) administered via the subcutaneous route into the left thigh and Simultaneous administration of Inactivated Hepatitis A vaccine, 0.5 mL liquid dose for intramuscular injection administered via the intramuscular route into the right thigh
  Interventions: Biological: Live attenuated chimeric Japanese Encephalitis vaccine; Biological: Inactivated Hepatitis A vaccine

INTERVENTIONS:
Biological: Live attenuated chimeric Japanese Encephalitis vaccine — 0.5 mL dose containing ≥ 4.0 log10 plaque forming units (PFU) administered via the subcutaneous route into the left thigh
  Other Names: Imojev
Biological: Inactivated Hepatitis A vaccine — 0.5 mL liquid dose for intramuscular injection administered via the intramuscular route into the right thigh
  Other Names: Havrix

SUMMARY:
This study was undertaken to assess the immunogenicity and safety of a booster dose of a live attenuated chimeric Japanese Encephalitis vaccine (JE-CV) after primary vaccination with SA14-14-2 in Thai children aged 1 to <5 years. In addition, to assess the impact of the duration interval after primary vaccination on subsequent booster response.

DETAILED DESCRIPTION:
The subject will receive one booster dose of IMOJEV with hepatitis A vaccine (inactivated vaccine of GlaxoSmithKline) as concomitant vaccine. Blood samples will be collected to assess for Japanese Encephalitis Neutralizing Antibody at baseline (pre-vaccination) and 4 week post -vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to <5 years on the day of inclusion
* History of received 1 dose of CD.JEVAX at 9-15 months prior to enrollment
* In good general health at the time of inclusion
* Provision of informed consent by the parent(s) or legal guardian(s)

Exclusion Criteria:

* Receipt of blood or blood products in the past 3 months
* Acute febrile illness on the day of vaccination (Body Temperature ≥ 38 ◦C)
* Previous receipt of 2 doses of any vaccine against JE virus
* Known hypersensitivity to any of the vaccine components
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Planned receipt of any live attenuated vaccine within 4 weeks following the trial vaccination

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kulkanya Chokephaibulkit, Professor, Principal Investigator — Siriraj Hospital

IPD SHARING:
Plan to Share IPD: No
The submission of study review and results to a peer-review journal is ongoing.

REFERENCES:
- [Derived] Sricharoenchai S, Lapphra K, Chuenkitmongkol S, Phongsamart W, Bouckenooghe A, Wittawatmongkol O, Rungmaitree S, Chokephaibulkit K. Immunogenicity of a Live Attenuated Chimeric Japanese Encephalitis Vaccine as a Booster Dose After Primary Vaccination With Live Attenuated SA14-14-2 Vaccine: A Phase IV Study in Thai Children. Pediatr Infect Dis J. 2017 Feb;36(2):e45-e47. doi: 10.1097/INF.0000000000001395. PMID 27846060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase IV study was conducted between 01 June 2014 and 04 July 2014 in accordance with ICH GCP. The study was approved by the Siriraj IRB. Written Informed Consent was obtained from all participants' parents or legal guardians before study entry.
Period: Overall Study
Arm/Group | Imojev
Started | 50
Completed | 49
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imojev
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: months] | 20.5 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Region of Enrollment [Number; unit: participants]
  Thailand | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Geometric Mean Titers Against the Japanese Encephalitis Chimeric Virus at 28 Days Post Vaccination
Description: Geometric mean titers were assessed using a Japanese encephalitis chimeric virus (JE-CV) 50% Plaque Reduction Neutralization Test (PRNT50).
Time Frame: Day 0 (Baseline) and Day 28 (post-vaccination)
Population: Per-protocol analysis
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Imojev
Number analyzed (Participants) | 49
titers | 9144 [7365 to 11353]

2. Secondary Outcome: Change From Baseline in Number of Participants With Seroprotection Against Japanese Encephalitis Chimeric Virus at 28 Days Post Vaccination
Description: Immunogenicity was assessed using a Japanese encephalitis chimeric virus (JE-CV) PRNT50 assay. Seroprotection was defined as the percentage of participants with a titer ≥10 (1/dil) at pre-vaccination and at Day 28 post-vaccination.
Time Frame: Day 0 (Baseline) and Day 28 (post-vaccination)
Measure: Number; unit: percentage of participants
Arm/Group | Imojev
Number analyzed (Participants) | 49
percentage of participants | 100

3. Secondary Outcome: Percentage of Number of Participants Reporting Immediate Reactions, Solicited Injection Site and Systemic Reactions, Unsolicited Adverse Events, and Serious Adverse Events Following Vaccination With IMOJEV™
Description: Immediate reactions: any reactions occurred within 30 minutes following vaccination; Solicited injection site reactions: Injection site Pain, Redness, and Swelling; Solicited systemic reactions: Fever (Temperature), Crying/Irritability, Drowsiness, Low Appetite and Skin Rash; Unsolicited adverse events: any adverse events spontaneously reported by participants regardless the causal relationship of adverse events to vaccine; Serious adverse events: Any adverse events that resulted in any of the following outcomes: death, a life threatening adverse event, in patient hospitalization or prolongation of existing hospitalization, a persistent or significant disability / incapacity, a congenital anomaly/birth defect, or any important medical events based upon appropriate medical judgment.
Time Frame: Up to 28 days post booster vaccination
Measure: Number; unit: percentage of participants
Arm/Group | Imojev
Number analyzed (Participants) | 49
percentage of participants
  Immediate reactions | 0
  Injection site pain | 10.2
  Injection site redness | 6.1
  Injection site swelling | 6.1
  Fever | 10.3
  Crying/Irritability | 8.3
  Drowsiness | 10.4
  Low Appetite | 8.2
  Skin Rash | 12.2
  Unsolicited adverse events | 49.0
  Serious adverse events | 0

ADVERSE EVENTS:
Time Frame: 28 days following vaccination
Description: Patients' parents/guardians were provided with rulers, digital thermometers, and diary cards to record daily temperature and any solicited local injection site reactions (pain, redness, and swelling) and general symptoms (fever, abnormal crying/irritability, drowsiness, loss of appetite and skin rash) during the 28-day period following each study vaccination. The occurrence of unsolicited (i.e. spontaneously reported) adverse events were recorded for up to 28 days following vaccination.
Arm/Group | Imojev
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 31/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imojev (N=49)
Immediate reactions (General disorders) | 0 (0) — Any reactions occurring within 30 minutes following vaccination
Solicited local reactions (Skin and subcutaneous tissue disorders) | 6 (11) — Solicited injection site reactions including pain, redness, swelling
Solicited systemic reactions (General disorders) | 12 (25) — Solicited systemic reactions including fever, crying/irritability, drowsiness, low appetite, skin rash
Unsolicited adverse events (General disorders) | 24 (34) — Unsolicited adverse events are the spontaneously reported adverse events by patients or patients' parents/guardians

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes